# The Pediatric Artificial Pancreas Automated Initialization trial (PEDAP-AI): A Pilot Study of AI Advisor-Driven Pump Initiation and Parameter Adaptation in Young Children with Type 1 Diabetes

Statistical Analysis Plan

Version 2.0

Corresponds to Version 5.0 of the Protocol

# Version History

| SAP<br>Version | Version Author Approver Date Revision Description | | Revision Description | Study Stage | Protocol<br>Version<br>4.0 | |
|---|---|---|---|---|---|---|
| 1.0 | | | Initial | Pre-Enrollment | | |
| 2.0 | Zachariah<br>Reed | Craig<br>Kollman | May 10,<br>2024 | Updated to<br>accommodate<br>protocol changes<br>regarding enrollment<br>of pump users;<br>corrected definition of<br>CGM-measured<br>hypoglycemic events | In progress | 5.0 |

I agree to the terms defined by the placement of mysignature in this schoon reent Author:

Craig Kollman

Senior Statistician (JCHR Director of Biostatistics): 

| John Statistician | I am electronically signing this document | 2024-05-10 09:55-04:00 |

I agree to the terms defined by the place 2024-05-10 11:28-04:00

JCHR Project Director:

Marc D Bretom 18 2024.05.10 09:28:57 -04000

# T ABLE OF CONTENTS

| 1 | Stı | udy Overview | 4 |
|---|---|---|---|
| 2 | Co | onsistency | 7 |
| 3 | Sta | atistical Hypotheses | 7 |
| 4 | Sa | mple Size | 7 |
| 5 | Ou | atcome Measures | 7 |
| | 5.1 | Safety Endpoints | 7 |
| | 5.2 | Efficacy Endpoints | 8 |
| | 5.3 | Analysis Datasets and Sensitivity Analyses | 9 |
| | 5.4 | CGMMetrics Calculations | 9 |
| | 5.5 | Calculation of InsulinMetrics | 10 |
| | 5.6<br>Grou | Calculation of CGM and Insulin Metrics for Comparison with the PEDAP Historical Compa | itrol |
| | 5.7 | Analysis Windows | 10 |
| 6 | Ar | nalysis | 10 |
| ( | 5.1 | Analysis of the Hierarchical Endpoints | 10 |
| ( | 5.2 | Analysis of Secondary Endpoints | 11 |
| | 6.2 | 2.1 Comparison with Baseline | 11 |
| | 6.2 | 2.2 Comparison with PEDAP Historical Control | 11 |
| ( | 5.3 | Analysis of Exploratory Endpoints | 11 |
| ( | 6.4 | Additional Tabulations and Plots | 12 |
| 7 | Sa | fety Analyses | 12 |
| 8 | Int | rervention Adherence | 12 |
| 9 | Pro | otocol Adherence and Retention | 12 |
| 10 | Ba | seline Descriptive Statistics | 13 |
| 11 | De | evice Issues | 13 |
| 12 | Pla | anned Interim Analyses | 13 |
| 13 | Su | bgroup Analyses | 13 |
| 14 | Mi | issing Data | 14 |
| 15 | Mι | ultiple Comparisons/Mltiplicity. | 14 |
| 16 | Re | ferences | 14 |

#### Study Overview I

This document outlines the statistical analyses to be performed for the PEDAP-AI study. The following table provides an overview.

Table I. Study Ove,n iew

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Ti tle | The Pediatric Artificial Pancreas Automated Initialization trial (PEDAP-AI): A Pilot Study of Al Advisor-DrivenPump Initiation and Parameter Adaptation in Young Children wilh Type I Diabetes |
| Pfecis | A single-armpilot study of Al Advisor-drivenat-homeclosed loop system initiation and parameter adaptation inyou1hage2 to <6 yearsold. |
| Inn ·stigational De,i c.e | Tandemt:slim X2wi1hControl-IQ and!:connect mobile application and DexcomG6 or G7 system,connected to WA cloud-based Physician Dashboard |
| Objectins | The objective of the study is to obtain safety data and exploratory glycemic control data will hinitiation and use of a closed loop control (CLC) system (t:slim X2 with Control-IQ Technology) inyoung children with initial selection of pump parameters and subsequent periodic parameter adjustment driven by an Al-based Advisor system over a 8-week period. |
| Study Design | In this single-armintervention trial, all participants will use the study system (pump and CGM) in closed-loop mode for 8 weeks. |
| Nnmber of Sites | -3 USclinical centers |
| End points | The key safety outcomes are adverseevents related to hypoglycemia and hyperglycemia, CGM-measuredtime spent below 54mg/dL, and CGM-measuredtime spent above 250mg/dL CGM-measuredendpoints will be tested against baseline for non-inferiority <b>Efficacv</b> Glycemicoutcomes including time in target range 70-180 mg/dL (TIR) and various other CGM measures of hypo- and hyperglycemia will be assessed and tested for superiority against baselineand a matched historical control population from the prior PEDAP study that didnot involve the use of any Al-driven pump parameters. |
| Population | <ol> <li>Ke.v Inclusion C1i.te-ria</li> <li>Clinical diagnosis based on investigator assessment, of type I diabetes for at least I month</li> <li>Familiarity and use of a carbohydrate ratio formeal boluses</li> <li>Age;;;2 and &lt;6 yearsold</li> <li>Using a Dexcom CGM at the time of enrollment, withuse on at least 21 out of the prior 28 days</li> <li>Living withoneor more parent/legal guardianknowledgeableabout emergency procedures forsevere hypoglycemia andable to contact emergency services and study staff.</li> <li>Parent/guardianhas a phonethat canrun the Tandem!: connect Mobile App (typically Android 10 or above or iOS 15 or above)</li> <li>Willingness to use the!: connect Mobile App as needed during the study andensure connectivity for a dataupload at least onceper day</li> <li>Investigator has confidence that the parent cansuccessfully operate all study devices and is capable of adhering to the protocob</li> <li>Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides Jisp ro (Humalog) or aspart (Novolog) during the study for participants using a study-provided Tandem pump during the study.</li> <li>Total daily insulindose (TDD) at least 5 U/day</li> <li>Rody weightat least 20 lbs</li> <li>Villinoness not to start any new non-insulin ducose-lowerine: aizent durine: the course</li> </ol> |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | of thetrial 13. Participant and parent(s)/guardian(s)willingness to participatein all training sessions as directed by study staff 14. Pared/guardian proficient in reading and writing English 15. Live in the United States, with no plans to move outside the United States during the study period |
| | Ke.y ExclusionCriteria |
| | <ol> <li>Concurrent useofany non-insulin glucose-lowering ageot (including GLP-1 agonists, Symlin, DPP-4 inluoitors, SGLT-2 inluoitors, sulfonylureas)</li> <li>Hemophilia or any otherbleedingdisorder</li> <li>History of &gt;1 severe hypoglycemiceventwithseizure or loss of consciousness in the last 3 months</li> <li>History of &gt;1 DKA eveot inthe last 6 monthsnot related to illness, infusion set failure, or initialdiagnosis</li> <li>History of chronic reoal disease or curreotly on hemodialysis</li> <li>History of adrenal insufficieocy</li> <li>Hypoth} oidismthat is not adequately treated in theopinion of the investigatro</li> <li>Use of oral or injectable steroidswithin the last8 weeks</li> <li>Known, ongoing adhesive intolerance</li> <li>Plans to receive bloodtransfusions or erythropaetin injection during the course of the study</li> <li>Acondition, which in the opinion of the investigator or designee, would put the participantor study at risk</li> <li>Participation inanother pharmaceutical or device trial at the time of enrollment or during the study</li> <li>Having immediate family members employed by Tandem Diabetes Care, Inc. or Dexcom, Inc., or having a direct supen, sor at place of employment who is also directly involvedinconducting the clinical trial (as a study investigato, recordinator, etc.); or ha, jng a first-degree relative who is directly involvedin conducting the</li> </ol> |
| SampleSiu | Up to 45 screened participants with the goal of at least 30 participants completing the study pump use period |
| Intern ntion | t:slim X2 with Control-IQ Technology and t:connectmobileapplication withmobile bolus capabilities and Study CGM |
| Participant Duation | -8 weeks |
| Study Duration (planned | -8 months from first eorollmeot until last participant , isi t |
| Protocol On ·ni ew/Synopsis | After consent is signed, eligibility will be assessed. Eligible participants Willproceed to the mainstudy described below. Initial pump parameter settings will be reviewed by clinical sitestaff after uploading baseline personal CGM and insulin data to a web-based Al-driven Advisor interfac. The Advisor Willsuggest pump parameter settings that the study investigatormay either accept unchanged or else overridebased on clinical judgment if there are any safety concerns. A study pump will be configured with the resulting parameter values, the participant will be pro, ded with the study pump and study CGM and other supplie, s and the participant will beginhome use of the pump. Visits• willoccur at 3 days and at I, 2, 4, and 6 weeks, with each, sit including siteupload of pump/CGM data to the Adviso interface to obtain recommended adjustments to pump parameters. As before, the study investigatormay either accept unchanged or else override based on clinical judgment if there are any safety concerns. A final study visit willoccur at 8 weeks, at which time the study participant will be transitioned back to preferred post-study insulin therapy. A follow-up safety visit willoccur 3 days after the final, sit toconfirm successful transition post-study insulin therapy. * All stul, visits may be conducted ei. The remotehvia teleconference or else in verson at |

| P ARTICIPANT AREA | DESCRIPTION |
|-------------------|-------------------|
| | the clinical site |

The following table provides an overview of the schedule of study visits, phone contacts, and key procedures.

Table 2. Schedule of Study Vi its and Procedures

| | Screenin1<br>Visit* | Baseline - Pump Initiation** | 3d | lw | lw | 4 w | 6w | 8w | 8w<br>+Jd |
|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | Х | | | | | | | | |
| Eligibility Assessme <b>n</b> | X | | | | | | | | |
| Medical history/<br>height/weight | х | | | | | | | | |
| Central lab HbAlc | | X | | | | | | | |
| Study pump training | | Х | | | | | | | |
| Upload devidata from home | | | Χ | Χ | Χ | Χ | X | X | |
| Review diabetes management, <b>AEs and medicatios</b> | | Х | Х | Х | Х | Х | X | X | X |
| Manual pump parameter adjustmentonly if safety issue | | | An | y schedu | led or ur | nschedul | ed visit | | |
| AI-driven pump parameter initiation/adjustment | - | Х | Х | Х | Х | Х | X | | |

<sup>•</sup> Allscreening visit pro es mustbe completed within 28 days of eConsent.

<sup>••</sup> All Pump initiation visit pro ures must be completed within IO daysof screening visit procedure completion.

# 1 2 Consistency

2 This SAP is consistent with the study protocol statistics chapter (version indicated on the title page).

## 3 Statistical Hypotheses

- 4 The primary outcomes for this study are safety outcomes: hypoglycemia and hyperglycemia measured by
- 5 adverse events and CGM. Statistical hypotheses are stated for the CGM-measured outcomes only.
- 6 CGM-measured percentage below 54 mg/dL and CGM-measured percentage above 250 mg/dL will be
- 7 tested for non-inferiority over an 8-week period.
- 8 The null/alternative hypotheses are:
- 9 Percentage below54 mgldL:
  - a. *Null Hypothesis*: The difference in mean CGM-measured % below 54 mg/dL between the 8 weeks follow-up and baseline is greater than or equal to +0.5% (non-inferiority).
    - b. *Alternative Hypothesis*: The difference in mean CGM-measured% below 54 mg/dL between the 8 weeks follow-up and baseline is less than +0.5%.

## 14 Percentage above 250 mgldL:

- a. *Null Hypothesis*: The difference in mean CGM-measured % above 250 mg/dL between the 8 weeks follow-up and baseline is greater than or equal to +3% (non-inferiority)
- b. *Alternative Hypothesis*: The difference in mean CGM-measured% above 250 mg/dL between the 8 weeks follow-up and baseline is less than +3%.

# 19 4 Sample Size

10

11

12

13

15

16

17

18

25

28 29

- The study has not been formally powered to test any a priori hypothesis. The goal is to have at least 30
- 21 participants complete the 8-week trial period. Some outcomes will be compared between these
- 22 participants and a sample of participants from the prior PEDAP study.
- 23 S Outcome Measures
- 5.1 Safety Endpoints
  - Severe Hypoglycemia (SH) events and SH event rate per 100 person-years
- Diabetic ketoacidosis (DKA) events and DKA event rate per 100 person-years
- Reportable hyperglycemia adverse events with or without ketosis
  - o Events related to the study device
  - o Events not related to the study device
- Reportable hypoglycemia adverse events that are not severe
- Number of calendar days with any ketone level:::1.0 mmol/L
- 32 Hierarchical Safety Endpoints
- CGM-Measured
- o % Time>250 mg/dL (non-inferiority)
- o % Time < 54 mg/dL (non-inferiority)

| <i>36</i> | <u>Additional Safety Endpoints</u> |
|---|---|
| 37 | Other serious adverse events |
| 38 | Any adverse event rate per 100 person-years |
| 39 | Adverse device effects (ADE) |
| 40 | • Serious adverse device events (SADE) |
| 41 | Unanticipatedadverse device effects (UADE) |
| 42 | 5.2 Efficacy Endpoints |
| 43 | Hierarchical E fficacy Endpoints /tested for superiority compared with baseline) |
| 44 | CGM-Measured |
| 45 | o % Timein range70-180 mg/dL |
| 46 | o Mean glucose |
| 47 | o % Time>250 mg/dL |
| 48 | o % Time < 70 mg/dL |
| 49 | o % Time < 54 mg/dL |
| 50 | Secondary Endpoints |
| 51 | CGM-Measured |
| 52 | o % Time in range 70-140 mg/dL |
| 53 | o % Time>180 mg/dL |
| 54 | o $\%$ Time $> 300$ mg/dL |
| 55 | o % Time<60 mg/dL |
| 56 | o Glucose standard deviation |
| 57 | o Glucose coefficient of variation |
| 58 | o High bloodglucose index (HBGI) |
| 59 | o Low blood glucoseindex (LBGI) |
| 60 | o Weekly hyperglycemiceventrate |
| 61 | o Weekly hypoglycemiceventrate |
| 62 | o Binary |
| 63 | • % Time in range 70-180 mg/dL improvement from baseline to 8 weeks:::5% |
| 64 | • % Time in range 70-180 mg/dL improvement from baseline to 8 weeks:::10 |
| 65 | • % Time in range 70-180 mg/dL $>$ 70% and% time $<$ 70 mg/dL $<$ 4% |
| 66 | • Insulin |
| 67 | o Total daily insulin (units/kg) |
| 68 | o Percentage of total insulin delivered via basal |

| <i>69</i> | Exploratory En | <u>idpoints</u> |
|---|---|---|
| 70 | <ul> <li>Insulir</li> </ul> | ı |
| 71 | 0 | Total daily basal insulin (units/kg) |
| 72 | 0 | Total daily bolus insulin (units/kg) |
| 73 | 0 | Total daily manual bolus (units/kg) |
| 74 | 0 | Total daily automated bolus(units/kg) |
| 75 | 0 | Number of manual insulin doses per day |
| 76 | 0 | Number of manual insulin doses with carb announcement per day |
| 77 | 0 | Average daily profilebasal rate divided by total daily insulin in percentage points |
| 78 | 0 | Average carbohydrate ratio daily profile (C:I) multiplied by total daily insulin |
| 79 | 0 | Average insulin sensitivity factor daily profile (G:I) multiplied by total daily insulin |
| 80 | 5.3 An | alysis Datasets and Sensitivity Analyses |
| 81<br>82<br>83 | | in included in analyses of CGM and insulin outcomes, participantsmust provide at least GMdata for each of the baseline and trial phase and spend at least 50% of the study period mode. |
| 84<br>85<br>86<br>87<br>88 | All participants who enroll in the PEDAP-AI study will be included in the safety analyses of endpoints that are not measured by CGM. Analyses will include all events that occur between enrollment and the 3-Day Post-Study Safety contact or the end of the 71st day after the date of the Closed Loop Initiation visit- whichever is earlier. For participants who do not complete the study, the date of the final contact will be used in place of the 3-Day Post-Study Safety contact date. | |
| 89 | 5.4 CC | GM Mehics Calculations |
| 90<br>91 | Baseline value<br>the Screening v | es for each CGM metric will be computed from the most recent 28 days of CGM data before visit. |
| 92<br>93<br>94<br>95 | the end of the d<br>Initiation visit | attment period, CGM metrics will be calculated from the beginning of study pump useuntil day before the 8-Week visit date or the end of the 59th day after the date of the Closed Loop whichever is earlier. For participants who do not complete the study, the date of the final cused in place of the 8-Week visit date. |
| 96<br>97<br>98<br>99<br>100 | below 54 mg/d<br>intervening val<br>defined as a m<br>2 sensor values | ared hypoglycemicevent is defined as 15 consecutive minutes with a sensor glucose value dL. At least 2 sensor values <54 mg/dL that are 15 or more minutes apart plusno lues :::54 mg/dL are required to define an event. The end of the hypoglycemic event is inimum of 15 consecutive minutes with a sensor glucose concentration :::70 mg/dL. At least :::70 mg/dL that are 15 or more minutes apart with no intervening values <70 mg/dL are fine the end of an event. |
| 102<br>103<br>104<br>105<br>106 | above 300 mg/<br>intervening va<br>defined as a m | ared hyperglycernicevent is defined as 90 consecutive minutes with a sensor glucosevalue /dL. At least 2 sensor values >300 mg/dL that are 90 or more minutes apart plus no lues \$300 mg/dL are required to define an event. The end of the hyperglycernicevent is inimum of 15consecutive minutes with a sensor glucose concentration ::,180 mg/dL. At values::,180 mg/dL that are 15 or more minutes apart with no intervening values >180 |

mg/dL are required to define the end of an event.

106

**107** 

| 108 | 5.5 Calculationoflnsulin Metlics |
|---|---|
| 109<br>110 | Insulin metrics for comparisons between baseline and follow-up describe the seven daysprior to the visits. |
| 111<br>112<br>113<br>114 | Baseline insulin metrics will usedata reported from the Diabetes Screening CRF. Insulin metrics will be calculatedat 8 weeks using Tandem pump data. Insulin pump dataon at least Sof7 days will be required to calculate insulin metrics. Weight will only be recordedat the Screeningvisit. All calculations of units/kg will use this weight, |
| 115<br>116 | 5.6 Calc ula tion of CGM and Insulin Metlics for Comparison with the PEDAP Histor ical Conti·ol Group |
| 117<br>118<br>119<br>120<br>121 | Results from this PEDAP-AI study will be compared with those from a sample of participants from the prior PEDAP study. For this analysis, participants from the prior PEDAP study will be limited to those whose RCT baseline HbAlc values are no more than 0.2 percentage points outside of the range observed among the PEDAP-AI participants. Basdine metrics for the PEDAP historical control group will be as reported for the PEDAP RCT. |
| 122<br>123<br>124<br>125<br>126<br>127<br>128<br>129<br>130<br>131 | The follow-up period for these comparisons will be the 7m and gm weeks of study pump use. For PEDAP-AI participa,ntsthis will be the period from the adjustment of pump settings at the 6-Week visit until the end of the day before the 8-Week visit. If the 6-Week visit is missed, data from the 14 days before the 8-Week visit will be used. PEDAP-AI participants will be excluded from these analyses if they miss the 8-Week visit. For the PEDAP historical control group, follow-up metrics will be calculated from the 14 daysprior to the 56m day after the date of the beginning of study pump use. These data will come from the RCT phase for those who were assigned to the CLC group and Extension phase for those who were assigned to the SC group. Participants must have spent at least SO% of the time between pump initiation and the end of the follow-up period in closed-loopmode, and provided at least 168 hours of data in both the baseline and follow-up periods for inclusion in analyses. |
| 132<br>133<br>134<br>135 | Baseline insulin metrics will usedata reported from the Diabetes Screening CRF. Insulin data must be present on at least 70% of follow-up days to calculate insulin metrics. The day of the 6-Week visit will be excluded from the calculation of PEDAP-AI participants' insulin metrics. Calculation of units/kg will use the weight from the Screening visit only. |
| 136 | 5.7 Analysis \Vindows |
| 137<br>138<br>139 | For any analysis or tabulation that involves HbAlc measured at the Closed Loop Initiation visit, the sample must be collected no earlier than three daysprior to the visit and no later than 21 days after the visit. |
| 140 | 6 Analysis |
| 141 | 6.1 Analysis of the Hiera rchical Endpoints |
| 142<br>143<br>144<br>145<br>146<br>147<br>148 | Summary statistics will be reported for the hierarchical endpoints at baseline and during follow-up as well as for differences from baseline. 24-hr profile plots will be drawn for follow-up. Boxplots will be drawn for baseline and follow-up. Scatter plots will be drawn for follow-up versus baseline. 95% confidence intervals will be constructed for the change from baseline to 8 weeks. For% <54 mg/dL and% >250 mg/dL, tests of non-inferioritywill be conducted using paired <i>t-tests</i> . The limits will be 0.5% for% <54 mg/dL and 3% for%>250mg/dL. If these outcomes are determined to be non-inferior, they will be tested for superiority in a hierarchy with% 70-180 mg/dL, mean gluco,se and% <70 mg/dL. Tests of |

superiority will be two-sided paired *t-tests*. If the distribution of changes is skewed then robust methods

will be used instead.

149

1SO

- To preserve the overall type 1 error among the formal comparisons, a hierarchy will be used in the following order:
   CGM % >250 mg/dL (non-inferiority; limit=3%)
   CGM % <54 mg/dL (non-inferiority; limit=0.5%)</li>
- CGM% 70-180mg/dL(superiority)
- Mean glucose (superiority)
- CGM% >250 mg/dL (superiority)
- CGM% < 70 mg/dL (superiority)
- CGM% <54 mg/dL (superiority)
- 160 If any of these comparisons result in a p-value >0.05, then formal testing will stop and p-values will not
- be generated for any subsequent testson the list. Note that the point estimates and confidence intervals
- will be generated for metrics regardless of statistical significance.

# 6.2 Analysis of Secondary Endpoints

# 6.2.1 Comparison with Baseline

- Summary statistics will be reported for baseline, follow-up, and difference from baseline. For all
- 166 continuous outcomes, boxplots will be drawn for baseline and follow-up and scatter plots will be drawn
- 167 for follow-up versus baseline. 24-hr profile plots will be drawn for continuous CGM-measured endpoints
- during follow-up.

163

164

175

184

- 169 Change over time will be compared with a paired *t-test* when the change appears approximately normal,
- and using robust methods when the change is skewed. Ninety-five percent confidence intervals of the
- 171 changes from baseline will be derived from these tests.
- For the binary outcome% time in range 70-180 mg/dL>70% and% time <70 mg/dL <4,% the
- proportion will be compared between baseline and follow-up with Barnard's exact test. A ninety-five
- percent confidence interval of the change from baseline will be derived from this test.

## 6.2.2 Comparison with PEDAP Hist01ical Control

- 176 Comparisons between the PEDAP-AI group and the PEDAP historical control group will be made for all
- of the hierarchical and secondary efficacy endpoints listed above. Continuous endpoints will be compared
- between the PEDAP-AI and PEDAP cohorts using a linear model adjusting for the baseline value age at
- initiation of closed loop use, use of pump or MDI before initiation of closed loop use and clinical center
- as fixed effects. Binary endpoints will be compared using a logistic model that adjusts for the same
- effects Summary statistics for baseline, follow-up, and change from baseline will be reported by study
- along with the adjusted differences between the studies and their 95% confidence intervals. Boxplots
- displaying baseline and follow-up for both groups will be drawn for continuous outcomes.

# 6.3 Analysis of Exploratory Endpoints

- Nop-valueswill be calculated for exploratory analyses. Summary statistics for total daily basal insulin
- and total daily bolus insulin will be tabulated for baseline, 8 weeks and change from baseline to 8 weeks.
- For all other outcomes, summary statistics will be tabulated for 8 weeks. Boxplots for the follow-up
- period will be drawn for all outcomes. Boxplots for baseline will be given for total daily basal insulin and
- total daily bolus insulin. Summary statistics for the final 2-week period will be displayed side-by-side
- with those of the PEDAP historical control group.

#### Additional Tabulations and Plots 191 6.4 192 Summary statistics will be tabulated by daytime (6 00 am - 9:59 pm) and nighttime (10:00 pm - 5:59 am) 193 during baseline and the 8 weeks of follow-up for each of the continuous CGM-measured outcomes listed 194 in 5.2. 195 During the trial period, the closed-loop system will include a periodic parameter adjustment driven by an 196 Al-based Advisor system. Tabulatio, ns 24-hour profile plo, ts and boxplots of the continuous CGMmeasured outcomes listed in 5.2 will be generated for each of thesix adaptation periods and the two 4-197 198 week periods of the study. 199 The end of the first 4-weekperiod will be the adjustment of pump settings at the 4-Week visit. The end of the second 4-weekperiod will be the end of the day before the 8-Week visit date or the end of the 59th day 200 after the date of the Closed Loop Initiation visit- which ever is earlier. This date will also serve as the end 201 202 of the sixth adaptation period, which will begin at the 6-Week visit. The other five adaptation periods will include data from the adjustment of pump settings at the visit until the adjustment of pump settings at the 203 subsequent visit. If the subsequent visit is missed or out-of-window, the end of the period will be the end 204 205 of the day on the latest date that would be in-window for the visit. If a participant misses a vi,sit they will be absent from the period begun by that visit. Participants must provide CGM data for at least 75% of the 206 time period to be included in the plots and tabulations for that time period. 207 208 7 Safe ty Analyses 209 Hierarchical safety endpoints will be analyzed according to the directions in 6.1. All safety endpoints listed in 5.1 will be summarized in tables. Details of each reportable adverse event will be provided in a 210 211 listing. 212 **Intervention Adherence** 8 213 The following will be tabulated for the 8-weekstudy period to assess intervention adherence: 214 PercenttimeofCGMsensoruse Percent time of closed-loop system use 215 Percent time in different operational modes 216 217 Percent of Al recommendations that are accepted without any study physician adjustments 218 For Al recommendations that are adjusted, tabulation of initial and adjusted values 219 System use metrics will be calculated from the beginning of study pump useuntil the end of the day 220 before the 8-Week visit date or the end of the 59th day after the date of the Closed Loop Initiation visitwhichever is earlier. For participants who do not complete the study these metrics will be prorated: the 221 date of the final contact will be used in place of the 8-Week visit date. 222 223

## **Protocol Adherence and Retention**

- The following tabulations and analyses will be performed to assess protocol adherence for the study: 224
- 225 Number of protocol and procedural deviations
- Flowchart accounting for all enrolled participants 226
- 227 Flowchart of all participants at all scheduled visits and phone contacts after treatment initiation
- 228 Number of and reasons for unscheduled visits and phone calls

| 229 | <ul> <li>Number of participants who stopped treabnent and reasons</li> </ul> |
|---|---|
| 230 | 10 Baselin e Desa i ptive Statistics |
| 231<br>232<br>233 | Baseline demographic and clinical characteristics of all participants included in the primary analysis will be summarized in a table using summary statistics appropriate to the distribution of each variable. Characteristics will include: |
| 234 | • Age |
| 235 | Diabetes duration |
| 236 | BMI percentile |
| 237 | • Sex |
| 238 | Race/ethnicity |
| 239 | Parents' highest education level |
| 240 | Annual householdincome |
| 241 | Health insurance |
| 242 | HbAlc at initiation of closed loop use |
| 243 | Insulin modality |
| 244 | Total daily insulin (units/kg) |
| 245 | <ul> <li>Number of injections of short-acting insulin per day</li> </ul> |
| 246 | • Number of diabetic ketoacidosis events in the past 12 months |
| 247 | • Number of severe hypoglycemia events in the past 12 months |
| 248 | 11 DeviceIssues |
| 249 | The following will be tabulated for the 8-week study period to assess device issues: |
| 250 | Device malfunctions requiring study team contact and other reported device issues |
| 251 | Rate of different failure events and alarms per 24 hours recorded by the Control-IQ system |
| <ul><li>252</li><li>253</li><li>254</li></ul> | Tabulations will include all events that occur between enrollment and the 3-Day Post-Study Safety contact or the end of the 71" day after the date of the Closed Loop Initiation visit- whichever is earlier. Details of device issues will be provided in a listing. |
| 255 | 12 Planned Inteli m An al yses |
| 256 | No formal interim efficacy analyses are planned. |
| 257 | The DSMB will review safety data at intervals, with no formal stopping rules. |
| 258 | 13 Subgroup Analyses |
| 259<br>260<br>261 | With only 30 participants, the ability to evaluate subgroups is limited. However, percentage of timespent >250 mg/dL and% of timespent <54 mg/dL over 8 weeks will be explored separately in baseline HbAlc, race/ethnici,ty MDI or pump use at enrollment, and sex. No p-values will be calculated for these analyses. |

- 262 14 Missing Data
- 263 All comparisons will be restricted to available cases.

# 264 15 Multiple Compalisons/Multiplicity

- 265 For the baseline versus follow-up comparisons of the metrics mentioned in 6.1, the overall type I error
- 266 will be preserved using the hierarchical procedure described above. For all other analyses the false
- 267 discovery rate will be controlled using the adaptive Benjamini-Hochberg procedure. The categories for
- 268 the FDR correction will be:
- Baseline vs follow-up for CGM-measured endpoints
- Baseline vs follow-up for insulin endpoints
- PEDAP-AI vs PEDAP for CGM-measured endpoints
- PEDAP-AI vs PEDAP for insulin endpoints

## 273 16 References

1. Benjamini Y, Hochberg Y. On the adaptive control of the false discovery rate in multiple testing with independent statistics. *Journal of Educational and Behavioral Statistics*. 2000;25(1):60-83.